CLINICAL TRIAL: NCT03310190
Title: Post-Marketing Observational Study (PMOS) to Describe the Management and the Use of Healthcare Resources in Patients With Chronic Lymphocytic Leukemia (CLL) Initiating Venetoclax in Routine Clinical Practice (DEVOTE)
Brief Title: Study to Describe the Management and the Use of Healthcare Resources in Patients With Chronic Lymphocytic Leukemia (CLL) Initiating Venetoclax in Routine Clinical Practice
Acronym: DEVOTE
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P16-489
Record Dates: First submitted 2017-10-11; First posted 2017-10-16 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia (CLL); Deletion of the short arm of chromosome 17 (Del[17p]); Relapse Chronic Lymphocytic Leukemia; Refractory Chronic Lymphocytic Leukemia; Chronic Lymphocytic Leukemia with deletion of the short arm of chromosome 17; Cancer
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Chromosome 17 deletion; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants receiving venetoclax: Participants with Chronic Lymphocytic Leukemia (CLL) receiving venetoclax.

SUMMARY:
A study to assess the real-life management and use of healthcare resources during the initiation of:

* Venetoclax in combination with rituximab is indicated for the treatment of adult participants with chronic lymphocytic leukemia (CLL) who have received at least one prior therapy.
* Venetoclax in participants with CLL with the deletion of the short arm of chromosome 17 (del[17p]) who have received at least 1 prior therapy or participants with CLL without del(17p) who have received at least 1 prior therapy and for whom there are no other available treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Patient's physician prescribed venetoclax as per product monograph independent of the patient participation in this study.
* Has chronic lymphocytic leukemia (CLL) and has received at least one prior therapy.

Exclusion Criteria:

* Currently participating in an interventional study.
* Has other condition that, in the opinion of the treating physician, prohibits the patient from participating in the study or obscures the assessment of the treatment of CLL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with Chronic Lymphocytic Leukemia (CLL) who have received at least one prior therapy
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Duration of Prophylactic Hospitalization | Up to approximately 6 weeks
  Duration of prophylactic hospitalization is defined as the date of discharge - the date of admission + 1.
Number of Hours from Dosing to Blood Draw | Baseline (Day 0)
  Number of hours between laboratory assessments and the first dose of each ramp-up dose for venetoclax
Intravenous (IV) fluid hydration | Up to 24 weeks after first dose of venetoclax
  Type of IV fluid participant was on hydration, rate and duration are assessed.
Percent of Participants with Tumor Burden of Low, Medium, and High | Baseline (Day 0)
  Percent of participants with tumor burden of low, medium, and high.
Other Actions Taken within the First 24 Hours of each Dose Ramp-up | Up to approximately 6 weeks
  Other actions taken within the first 24 hours of each dose ramp-up, for example, prophylaxis treatment
Change from Baseline in Health Care Resource Utilization (HCRU) | Up to 24 weeks after first dose of venetoclax
  HCRU will be evaluated using self-administered questionnaire aimed at measuring the patient's health care resource utilization.
Change in Metabolites Post Dose | Up to 24 weeks after first dose of venetoclax
  Change in metabolites (potassium, creatinine, uric acid, phosphorus, calcium) post dose.
Percentage of Participants with Prophylactic Hospitalization | Up to approximately 6 weeks
  Percentage of participants with prophylactic hospitalization is defined as the percentage of participants who are hospitalized for prophylactic measures.
Reasons for Dose Interruptions | Up to 24 weeks after first dose of venetoclax
  Reasons for dose interruptions.
Change in Creatinine Clearance | Up to 24 weeks after first dose of venetoclax
  Change in creatinine clearance is defined as the change of creatinine clearance from Baseline (Day 0).
Number of Hours for Dose Interruptions | Up to 24 weeks after first dose of venetoclax
  Number of hours for dose interruptions is defined as the duration of dose interruptions in hours. If more than one does interruption occurs, the total number of hours for dose interruption will be calculated.
Number of Weeks for Ramping up Venetoclax Dose to 400 mg daily (QD) or maximum dose reached | Up to approximately 6 weeks
  Number of weeks for ramping up to Venetoclax 400 mg QD or maximum dose reached as the duration of the ramping-up period in weeks.
Number of Days on Each Dose of Venetoclax | Up to 24 weeks after first dose of venetoclax
  Number of days on each dose of venetoclax is defined as the date of first exposure to the dose - the date of the last exposure to the dose + 1.

SECONDARY OUTCOMES:
Percentage of Participants with Other Mutations | Baseline (Day 0)
  Percentage of participants with other mutations.
Weeks since Last CLL Relapse | Baseline (Day 0)
  Duration of time from most recent CLL relapse and Baseline (Day 0).
Percentage of Participants with Major Co-Morbidities | Baseline (Day 0)
  Percentage of participants with major co-morbidities including medical history/surgery and transplant prior to Baseline (Day 0).
Percentage of Participants with Exposure to Ibrutinib and/or Idelalisib Prior to Baseline | Baseline (Day 0)
  Participants with previous exposure to ibrutinib and/or idelalisib prior to Baseline (Day 0).
Change from Baseline in EORTC QLQ-C30 Scores | Up to 24 weeks after first dose of venetoclax
  Change from baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) scores.
Change from Baseline in Eastern Cooperative Oncology Group Performance Status | Up to 24 weeks after first dose of venetoclax
  Change from baseline in Eastern Cooperative Oncology Group (ECOG) performance status.
Change from Baseline in QLQ-CLL17 Scores | Up to 24 weeks after first dose of venetoclax
  Change from baseline in Quality of Life Questionnaire - Chronic Lymphocytic Leukemia (QLQ-CLL)17 scores.
Weeks Since Initiating First Line of Therapy for CLL | Baseline (Day 0)
  Duration of time in weeks from date of first line of therapy administered for CLL to Baseline (Day 0).
Percent of Participants at Each Stage in the Rai Staging System | Baseline (Day 0)
  Percent of participants at each stage in the Rai Staging System for CLL.
Percentage of Participants with Del(17p) | Baseline (Day 0)
  Percentage of participants with the deletion of the short arm of chromosome 17 (Del[17p]).
Percent of Participants at Each Stage in the Binet Staging System | Baseline (Day 0)
  Percent of participants at each stage in the Binet Staging System for CLL.
Number of Prior Lines of Therapy for CLL | Baseline (Day 0)
  Number of prior lines of therapy for CLL before initiating administration with venetoclax.
Years to Treatment from Initial Diagnosis of Chronic Lymphocytic Leukemia (CLL) | Baseline (Day 0)
  Years to treatment with venetoclax (Baseline, Day 0) from initial diagnosis of CLL.
Weeks since the Last Line of Therapy (Agent) for CLL Prior to Baseline | Baseline (Day 0)
  Duration of time in weeks since line of therapy (agent) administered for CLL prior to Baseline (Day 0).
Weeks since First CLL Relapse | Baseline (Day 0)
  Duration of time in weeks from diagnosis of CLL to first relapse.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (13):
- Canada (13):
  - University of Calgary /ID# 166416, Calgary, Alberta
  - Cross Cancer Institute /ID# 166417, Edmonton, Alberta
  - Jack Ady Cancer Centre /ID# 217491, Lethbridge, Alberta
  - CancerCare Manitoba /ID# 170751, Winnipeg, Manitoba
  - The Moncton Hospital /ID# 166043, Moncton, New Brunswick
  - QE II Health Sciences Centre /ID# 213548, Halifax, Nova Scotia
  - William Osler Health System /ID# 202049, Brampton, Ontario
  - Health Sciences North /ID# 205817, Greater Sudbury, Ontario
  - Kingston Health Sciences Centre /ID# 169252, Kingston, Ontario
  - Ottawa Hospital Research Institute /ID# 166041, Ottawa, Ontario
  - Thunder Bay Regional Research Institute /ID# 204740, Thunder Bay, Ontario
  - Jewish General Hospital /ID# 166418, Montreal, Quebec
  - CISSSBSL -Hopital regional de Rimouski /ID# 201202, Rimouski, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=P16-489&Latitude=&Longitude=&LocationName=#additional-resources-section